CLINICAL TRIAL: NCT06073093
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled, Dose-ranging, Efficacy and Safety Study of SAR441566 Plus Methotrexate in Adults With ModeratetoSevere Rheumatoid Arthritis
Brief Title: A Study to Evaluate SAR441566 Efficacy and Safety in Adults With Rheumatoid Arthritis
Acronym: SPECIFI-RA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRI17821; U1111-1288-8641 (Registry Identifier: ICTRP); 2023-503910-60-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- SAR441566 dose regimen A (Experimental): Participant will receive dose regimen A of SAR441566 for 12 weeks
  Interventions: Drug: SAR441566
- SAR441566 dose regimen B (Experimental): Participant will receive dose regimen B of SAR441566 for 12 weeks
  Interventions: Drug: SAR441566
- SAR441566 dose regimen C (Experimental): Participant will receive dose regimen C of SAR441566 for 12 weeks
  Interventions: Drug: SAR441566
- SAR441566 dose regimen D (Experimental): Participant will receive dose regimen D of SAR441566 for 12 weeks
  Interventions: Drug: SAR441566
- Placebo (Placebo Comparator): Participant will receive SAR441566-matching placebo for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR441566 — Tablet
  Arms: SAR441566 dose regimen A; SAR441566 dose regimen B; SAR441566 dose regimen C; SAR441566 dose regimen D
Drug: Placebo — Tablet
  Arms: Placebo

SUMMARY:
This is a parallel group, Phase 2, randomized, double-blind, placebo controlled, 5-arm, international, multicenter, 12-week proof of concept, dose finding study. It is designed to assess efficacy and safety of treatment with SAR441566 for 12 weeks. It will be conducted in male and female adult participants with moderate-to-severe rheumatoid arthritis (RA) not adequately controlled on methotrexate (MTX) and biologic/targeted synthetic disease modifying anti-rheumatic drug (DMARD) naive.

Study treatment includes investigational medicinal product (IMP: SAR441566 or placebo) added-on to a background therapy of MTX.

Study details include a run-in period (4 to 6 weeks) before randomization to determine eligibility, a treatment period (12 weeks ± 3 days) and a post-treatment period (safety follow-up) (2 weeks ± 3 days). The total number of scheduled study visits will be 8.

DETAILED DESCRIPTION:
The overall study duration for each participant will be approximately up to 149 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adult-onset RA classified by ACR/EULAR 2010 revised classification criteria for RA of at least 3 months duration, with the onset of signs and symptoms of RA of at least 6 months duration
* Moderate-to-severely active RA, defined as:

  * persistently active disease >= 6 tender and >= 6 swollen joints
  * high sensitivity C-reactive protein ≥ 4 mg/L
* Continuous treatment with MTX for at least 12 consecutive weeks prior to randomization and with stable dose/means of administration at least 6 weeks prior to the screening visit

  * MTX - 10 to 25 mg/week (or per local labeling requirements for the treatment of RA if the dose range differs) and folic/folinic acid (as part of MTX regimen)
* Inadequate clinical response to MTX at a dose of 10-25 mg/week after proper dose escalation according to local standards
* BMI within the range [18 - 35] kg/m^2 (inclusive)

Exclusion Criteria:

* Immunologic disorder other than RA, with the exception of secondary Sjogren's syndrome associated with RA, and medically controlled diabetes or thyroid disorder as per Investigator's judgement
* Any condition (other than RA) requiring oral, intravenous, IM, or intra-articular glucocorticoid therapy
* Uncontrolled polymyalgia rheumatica or fibromyalgia
* History of recurrent or recent serious infection (eg, pneumonia, septicemia) or infection(s) requiring hospitalization or treatment with IV anti-infectives (antibiotics, antivirals, antifungals, antihelminthics) within 30 days prior to D1. Infections(s) requiring oral anti-infectives (antibiotics, antivirals, antifungals, antihelminthics) within 14 days prior to D1
* Known history of or suspected significant current immunosuppression, including history of invasive opportunistic or helminthic infections despite infection resolution or otherwise recurrent infections of abnormal frequency or prolonged duration
* History of moderate-to-severe congestive heart failure (NYHA Class III or IV), recent cerebrovascular accident, or any other condition in the opinion of the Investigator that would put the participant at risk by participation in the protocol
* History of solid organ transplant
* History of alcohol or drug abuse within the past 2 years
* History of diagnosis of demyelinating disease such as but not limited to:

  * Multiple Sclerosis
  * Acute Disseminated Encephalomyelitis
  * Balo's Disease (Concentric Sclerosis)
  * Charcot-Marie-Tooth Disease
  * Guillain-Barre Syndrome
  * human T-lymphotropic virus 1 Associated Myelopathy
  * Neuromyelitis Optica (Devic's Disease)
* Planned surgery during the treatment period
* Participants who are Steinbrocker class IV functional capacity (incapacitated, largely or wholly bed-ridden or confined to a wheelchair, with little or no self-care)
* Vaccination with live or live-attenuated virus vaccine within 3 months prior to screening or plan to receive one during the trial including at least 3 months after the last dose of study drug
* Any non-live vaccine (eg, COVID-19) within 14 days prior to randomization or plan to receive one during the trial
* Participant with personal or family history of long QT syndrome
* Active malignancy, lymphoproliferative disease, or malignancy in remission for less than 5 years, except adequately treated (cured) localized carcinoma in situ of the cervix or ductal breast, or squamous cell carcinoma, or basal cell carcinoma of the skin
* Previous or current use of biologic therapy or targeted synthetic disease modifying anti-rheumatic drugs (tsDMARD - such as JAK inhibitors) for RA
* Use of oral glucocorticoid greater than prednisone 10 mg per day or equivalent per day, or a change in dosage within 4 weeks prior to screening. The dose of oral glucocorticoid must remain stable.
* Use of parenteral glucocorticoids or intra-articular glucocorticoids within 4 weeks prior to screening
* Initiation or change in dose for nonsteroidal anti-inflammatory drugs (NSAIDs) within 1 week prior to screening

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving at least 20% improvement from baseline in the American College of Rheumatology (ACR) score at week 12 | Baseline to Week 12
  ACR20 response criteria is a dichotomous composite endpoint indicating the proportion of participants with at least 20 percent improvement in the number of tender and swollen joints, and in three out of the remaining five ACR core-set measures: patient pain (VAS, No pain to Severe Pain), Patient Global Assessment of disease activity (VAS, Very well to Very Poor), physician global assessment of disease activity (VAS, Very good to Very bad), physical functioning assessment (Health Assessment Questionnaire-Disability Index [HAQ-DI]), and acute phase reactants (ESR or CRP mg/dl; in this study CRP will be used). ACR response is scored as a percentage improvement, comparing disease activity at two discrete time points. ACR20 is ≥ 20% improvement.

SECONDARY OUTCOMES:
Change from baseline in Disease activity score - C-reactive protein (DAS-28 CRP) at week 12 | Baseline to Week 12
  The DAS28-CRP is a composite endpoint. DAS28-CRP is comprised of clinical assessment of 28 swollen joint count (SJC)/ tender joint count (TJC), patient assessment of global disease activity and CRP mg/dL. It is a continuous measure allowing for measurement of absolute change in disease burden and percentage improvement.
  The DAS28 can be calculated using the following formula:
  DAS28 = 0.56 x 28TJC + 0.28 x 28SJC + 0.36 x Log(CRP+1) + 0.014 x GH + 0.96 The DAS28 provides a number indicating the current activity of the RA. A DAS28 above 5.1 means high disease activity, whereas a DAS28 below 3.2 indicates low disease activity and a DAS28 below 2.6 means disease remission.
Proportion of participants achieving at least 50% improvement from baseline in the ACR score at week 12 | Baseline to week 12
  ACR response is scored as a percentage improvement, comparing disease activity at two discrete time points. ACR50 is ≥ 50% improvement. ACR50 responders include ACR20 responders
Number of participants with Treatment-Emergent Adverse Events (TEAEs), serious AEs (SAEs), and AEs of special interest (AESIs) | Baseline to week 14
  Incidence of TEAEs, SAEs, and AESIs
Plasma pre-dose concentrations of SAR441566 | Week 2 to week 12
Plasma post-dose concentrations of SAR441566 | Week 0 to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (101):
- United States (17):
  - Amicis Research Center - Northridge - Nordhoff Street- Site Number : 8400023, Northridge, California
  - Inland Rheumatology & Osteoporosis Medical Group- Site Number : 8400004, Upland, California
  - UF Health Deerwood Park- Site Number : 8400020, Jacksonville, Florida
  - Life Clinical Trials- Site Number : 8400028, Margate, Florida
  - Future Care Solution - Miami- Site Number : 8400019, Miami, Florida
  - Innovia Research Center, Inc- Site Number : 8400026, Miramar, Florida
  - Integral Rheumatology and Immunology Specialists- Site Number : 8400010, Plantation, Florida
  - Clinical Research of West Florida - Tampa - North Howard Avenue- Site Number : 8400017, Tampa, Florida
  - Inspire Santa Fe Medical Group- Site Number : 8400029, Santa Fe, New Mexico
  - Arthritis and Osteoporosis Consultants of the Carolinas- Site Number : 8400012, Charlotte, North Carolina
  - Carolina Specialty Care- Site Number : 8400007, Statesville, North Carolina
  - Altoona Center for Clinical Research- Site Number : 8400002, Duncansville, Pennsylvania
  - Low Country Rheumatology- Site Number : 8400018, Summerville, South Carolina
  - American Indian Clinical Trials Research Network - Rapid City- Site Number : 8400022, Rapid City, South Dakota
  - Prolato Clinical Research Center- Site Number : 8400021, Houston, Texas
  - AARA Clinical Research - Lone Star Arthritis & Rheumatology Associates - Irving- Site Number : 8400031, Irving, Texas
  - Perceptive Pharma Research- Site Number : 8400009, Richmond, Texas
- Argentina (7):
  - Investigational Site Number : 0320005, Berazategui, Buenos Aires
  - Investigational Site Number : 0320004, Buenos Aires, Buenos Aires F.D.
  - Investigational Site Number : 0320001, Buenos Aires, Buenos Aires F.D.
  - Investigational Site Number : 0320003, Buenos Aires
  - Investigational Site Number : 0320007, Buenos Aires
  - Investigational Site Number : 0320006, Mar del Plata
  - Investigational Site Number : 0320002, San Miguel de Tucumán
- Brazil (5):
  - Centro Mineiro de Pesquisa- Site Number : 0760003, Juiz de Fora, Minas Gerais
  - Centro de Estudos em Terapias Inovadoras- Site Number : 0760004, Curitiba, Paraná
  - Hospital São Lucas Copacabana- Site Number : 0760007, Rio de Janeiro
  - CCBR / IBPClin - Instituto Brasil de Pesquisa Clínica- Site Number : 0760005, Rio de Janeiro
  - Centro Paulista de Investigaçăo Clínica - CEPIC- Site Number : 0760001, São Paulo
- Canada (4):
  - Investigational Site Number : 1240006, Calgary, Alberta
  - Investigational Site Number : 1240001, Brampton, Ontario
  - Investigational Site Number : 1240004, Windsor, Ontario
  - Investigational Site Number : 1240002, Sherbrooke, Quebec
- Chile (9):
  - Investigational Site Number : 1520001, La Serena, Coquimbo Region
  - Investigational Site Number : 1520003, Osorno, Los Lagos Region
  - Investigational Site Number : 1520005, Valdivia, Los Ríos Region
  - Investigational Site Number : 1520002, Talca, Maule Region
  - Investigational Site Number : 1520004, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520006, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520008, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520007, Viña del Mar, Región de Valparaíso
  - Investigational Site Number : 1520009, Santiago
- China (3):
  - Investigational Site Number : 1560004, Chengdu
  - Investigational Site Number : 1560003, Hefei
  - Investigational Site Number : 1560001, Shanghai
- Czechia (5):
  - Investigational Site Number : 2030006, Brno
  - Investigational Site Number : 2030002, Ostrava
  - Investigational Site Number : 2030008, Pardubice
  - Investigational Site Number : 2030001, Prague
  - Investigational Site Number : 2030003, Uherské Hradiště
- Investigational Site Number : 2680001, Tbilisi, Georgia
- Germany (3):
  - Investigational Site Number : 2760002, Berlin
  - Investigational Site Number : 2760001, Hamburg
  - Investigational Site Number : 2760003, Ratingen
- Greece (3):
  - Investigational Site Number : 3000001, Athens
  - Investigational Site Number : 3000002, Heraklion
  - Investigational Site Number : 3000003, Thessaloniki
- India (7):
  - Investigational Site Number : 3560006, Ahmedabad
  - Investigational Site Number : 3560002, Bengaluru
  - Investigational Site Number : 3560001, Chennai
  - Investigational Site Number : 3560010, Hyderabad
  - Investigational Site Number : 3560007, Kolkata
  - Investigational Site Number : 3560011, Nashik
  - Investigational Site Number : 3560005, Surat
- Japan (10):
  - Investigational Site Number : 3920005, Nagoya, Aichi-ken
  - Investigational Site Number : 3920007, Kamogawa, Chiba
  - Investigational Site Number : 3920006, Sapporo, Hokkaido
  - Investigational Site Number : 3920009, Sapporo, Hokkaido
  - Investigational Site Number : 3920004, Kawachi-Nagano, Osaka
  - Investigational Site Number : 3920003, Toyonaka, Osaka
  - Investigational Site Number : 3920002, Fuchū, Tokyo
  - Investigational Site Number : 3920008, Nagasaki
  - Investigational Site Number : 3920011, Tokorozawa
  - Investigational Site Number : 3920001, Toyota
- Investigational Site Number : 4800001, Vacoas, Mauritius
- Mexico (3):
  - Investigational Site Number : 4840002, Mexico City, Mexico City
  - Investigational Site Number : 4840001, Chihuahua City
  - Investigational Site Number : 4840003, Mérida
- Poland (6):
  - Investigational Site Number : 6160004, Poznan, Greater Poland Voivodeship
  - Investigational Site Number : 6160001, Lublin, Lubusz Voivodeship
  - Investigational Site Number : 6160002, Lublin, Lubusz Voivodeship
  - Investigational Site Number : 6160003, Bialystok, Podlaskie Voivodeship
  - Investigational Site Number : 6160005, Bytom, Silesian Voivodeship
  - Investigational Site Number : 6160006, Grodzisk Mazowiecki
- Caribbean Medical Research Center- Site Number : 8400027, San Juan, Puerto Rico
- Slovakia (2):
  - Investigational Site Number : 7030003, Nové Mesto nad Váhom
  - Investigational Site Number : 7030001, Piešťany
- South Africa (6):
  - Investigational Site Number : 7100002, Cape Town
  - Investigational Site Number : 7100003, Cape Town
  - Investigational Site Number : 7100001, Pretoria
  - Investigational Site Number : 7100005, Pretoria
  - Investigational Site Number : 7100004, Pretoria
  - Investigational Site Number : 7100007, Stellenbosch
- Spain (8):
  - Investigational Site Number : 7240001, A Coruña, A Coruña [La Coruña]
  - Investigational Site Number : 7240002, Santiago de Compostela, A Coruña [La Coruña]
  - Investigational Site Number : 7240006, Santiago de Compostela, A Coruña [La Coruña]
  - Investigational Site Number : 7240005, Seville, Andalusia
  - Investigational Site Number : 7240004, Sabadell, Castille and León
  - Investigational Site Number : 7240008, Chiclana de la Frontera
  - Investigational Site Number : 7240007, Madrid
  - Investigational Site Number : 7240003, Málaga

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org